CLINICAL TRIAL: NCT02614820
Title: The Safety, Efficacy and Tolerability of Remote Ischemic Preconditioning as a Therapy to DMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JZheng
Record Dates: First submitted 2015-11-17; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Ischemic preconditioning; sefety; efficacy; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- treatment group (Experimental): inflation of a blood pressure cuff on the bilateral thighs to 150 mm Hg for four 5-minute intervals
  Interventions: Procedure: Remote Ischemic Preconditioning Training Apparatus
- control group (Other): inflation of a blood pressure cuff on the bilateral thighs to 40 mm Hg for four 5-minute intervals
  Interventions: Procedure: Remote Ischemic Preconditioning Training Apparatus

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning Training Apparatus

SUMMARY:
Background: Duchenne muscular dystrophy (DMD) is an X chromosome recessive hereditary disease and mainly characterized by progressive muscle weakness and atrophy. Glucocorticoid is the only proven effective medicine,while side effects limit its use. Recent studies have shown that the vascular density in the DMD patients' muscle is decreased,so muscle are in ischemic and anoxic. Remote ischemic preconditioning(RIPC) can improve the capable of resistanting ischemia and hypoxia and maybe a potential therapy for DMD patients.

Methods: 100 patients (aged 2 to 6 years)will be divided into two groups(treatment and control groups) randomly. Treatment group will receive an RIPC stimulus (inflation of a blood pressure cuff on the bilateral thighs to 150 mm Hg for four 5-minute intervals) while control group will receive a similar stimulus (inflation of a blood pressure cuff on the bilateral thighs to 40 mm Hg for four 5-minute intervals). Serum kinase level ,Blood levels of myoglobin, Evaluation of motor function(Four steps test;6-minute walking test) and MRI of lower limbs）at 0 days, 3 days, 3months ,6months.

Purpose：

1. To evaluate the safety and tolerability of remote ischemic preconditioning for DMD patients
2. To identify the effectiveness of remote ischemic preconditioning for DMD patients.

ELIGIBILITY:
Inclusion Criteria:Genetic analysis of DMD; from 2 to 6 years old ;without other diseases .

-

Exclusion Criteria: other congenital diseases;upper respiratory infection, gastroenteritis, vaccination, trauma.

-

Ages: 2 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Serum CK value | 0 day
Serum CK value | 3 days
Serum CK value | 3 months
Serum CK value | 6 months
Serum myoglobin values | 0 day
Serum myoglobin values | 3 days

SECONDARY OUTCOMES:
Serum myoglobin values | 3 months

OTHER OUTCOMES:
Serum myoglobin values | 6 months
6-minute walking test | 0 day
6-minute walking test | 3 days
6-minute walking test | 3 months
6-minute walking test | 6 months
T2 values | 0 day
T2 values | 3 days
T2 values | 3 months
T2 values | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shiwen wu, Beijing, China